CLINICAL TRIAL: NCT03901495
Title: Differential Diagnosis Assessment in Ambulatory Care With an Automated Medical History-Taking Device: A Confirmatory Pseudo-Randomized Study
Brief Title: DD Assessment With Diaana #2
Acronym: DiaanaRCT#2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adrien Schwitzguebel (Other)
Responsible Party: Sponsor-Investigator, Adrien Schwitzguebel, Principal investigator, Independant physician, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UNIGE_Diaana
Record Dates: First submitted 2019-03-02; First posted 2019-04-03 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Decision Making; Computer-assisted; General Practitioners; Patient Engagement
Keywords: differential diagnosis; hospital outpatient clinics; clinical applications software
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Masking Description: The first 50 eligible patients of the emergency outpatient unit in Geneva University Hospital are recruited into the control group (without access to "Diaana"). The next 50 eligible patients are recruited into the intervention group (with access to "Diaana").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaana (Experimental): 1. The patient fullfill Diaana
  2. The resident physician takes connaissance of the Diaana summary
  3. The resident physician see the patient in consultation. He establishes his DD without having access to the complementay exams (blood tests, x-ray, ...)
  4. The senior physician see the patient in consultation. He establishes his DD without having access to the complementay exams (blood tests, x-ray, ...)
  Interventions: Other: Diaana
- Control (No Intervention): 1. The resident physician see the patient in consultation. He establishes his DD without having access to the complementay exams (blood tests, x-ray, ...)
  2. The senior physician see the patient in consultation. He establishes his DD without having access to the complementay exams (blood tests, x-ray, ...)

INTERVENTIONS:
Other: Diaana — Diaana, the AMHTD used, functions as follows: on the basis of an interactive questionnaire completed by the patient before the consultation, it performs an exhaustive anamnesis focused on the problem and proposes a panel of DDs with a high sensitivity. The artificial reasoning system of "Diaana" mimics how a specialist physician would reason to establish a DD. The information transmitted is in an easy-to-use form for the physician that includes a summary of the anamnesis centered on relevant elements from the questionnaire and a list of possible diagnoses with their emergency level, potential contributing factors, and first-line management proposals.
  Other Names: Automated medical history-taking device (AMHTD)
  Arms: Diaana

SUMMARY:
Single-center, unblinded, 1:1 parallel pseudo-randomized efficacy trial.

In the intervention group only, resident physicians will be assisted by the automated medical history-taking device "Diaana" during their consultations in outpatient ambulatory unit of the Geneva University Hospital.

In both groups, the differential diagnosis of the resident physician will be compared to the gold-standard differential diagnosis of the senior physician.

DETAILED DESCRIPTION:
Automated medical history-taking devices (AMHTD) are emerging tools with the potential to increase the quality of medical consultations by providing physicians with an exhaustive, high-quality, standardized anamnesis and differential diagnosis. In this study, the investigators aimed to establish whether an AMHTD of interest, "Diaana", allowed the physician to establish a more precise differential diagnosis.

A single-center, unblinded, 1:1 parallel pseudo-randomized efficacy trial will be performed. No follow-up is necessary, because patients are seen once and all data are collected on this time. The study will take place in the emergency outpatient unit of Geneva University Hospital and include patients suffering from symptoms covered by Diaana.

Patients in the intervention group will fullfil Dianna. Then, the resident physician will read Diaana summary, perform his consultation, and fullfil case report form, including his differential diagnosis. Then, the senior physician will see the patient and establish the gold-standard differential diagnosis. In the control group, the residents will directely establish a differential diagnosis, without the help of Diaana.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency outpatient unit of Geneva University Hospital
* Patients suffering from symptoms localized to the superior or inferior member, the back, hand the chest wall.

Exclusion Criteria:

* Strictly dermatologic concerns
* Toes and inversion ankle trauma (because the diagnosis of those conditions is generally obvious)
* Medical condition considered as urgent
* Inability to complete de digilatized Diaana form (sight problems, language, inability to use a tablet computer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Differential diagnosis established by the resident physician | At day 0
  The resident physician will select up to 5 diagnose in an exhaustive list. The senior physician will do the same in order to establish the gold-standard differential diagnosis.
  The accuracy of the resident's differential diagnosis will be measured as the percentage of correct diagnose selected by the resident compared to the gold standard.

SECONDARY OUTCOMES:
Consultation time | At day 0
  The resident's consultation (with and without the patient) will be measured by the research coordinator. Consultation time will be compared between groups. A shorter consultation time will be considered as a better outcome.
Patient satisfaction | At day 0
  Into the experimental group, the patient's satisfaction will be evalued on a Lickert 1-4 scale. 1= fully dissatisfied; 2 = partially dissatisfied; 3 = partially satisfied; 4 = fully satisfied
Differential diagnosis estabished by Diaana | At day 0
  The Diaana system will select diagnoses in an exhaustive list. The senior physician will select up to 5 diagnose in an exhaustive list in order to establish the gold-standard differential diagnosis.
  The accuracy of the differential diagnosis established by the Diaana system will be measured as the percentage of correct diagnose selected compared to the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Spechbach, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes measures will be made avaliable
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: Data will be avaliable within 3 months of the study completion
Access Criteria: Under request to the sponsor.

REFERENCES:
- [Derived] Healey B, Schwitzguebel A, Spechbach H. Differential Diagnosis Assessment in Ambulatory Care With a Digital Health History Device: Pseudorandomized Study. JMIR Form Res. 2025 Oct 1;9:e56384. doi: 10.2196/56384. PMID 40205939